CLINICAL TRIAL: NCT06859528
Title: Step Up to PD: A Community-based Walking Program for People With Parkinson's Disease
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: St. Louis University (Other)
Responsible Party: Principal Investigator, Jason Longhurst, Assistant Professor, St. Louis University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 34235
Record Dates: First submitted 2025-02-27; First posted 2025-03-05 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Parkinson Disease; Parkinson Disease, Idiopathic
Keywords: Walking; Physical Activity; Social Connectedness; Loneliness
MeSH Terms: conditions — Parkinson Disease; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Attend group community walking program for 60 minutes each week (Experimental): Participants will participate in one, 60-minute group walk using Nordic poles at the Missouri Botanical Gardens for at least 6 months, with an optional continuation upto 12 months. Participants will be assessed before the program begins, after 6-months, and after 12 months. Falls will be prospectively collected for 6 months following completion of the program.
  Interventions: Behavioral: Community Walking Program

INTERVENTIONS:
Behavioral: Community Walking Program — This is a group, community walking program at local parks using Nordic walking poles. Participants will be encouraged to walk briskly but safely for 60 minutes one time per week with the ultimate goal of using this community walking program to drive behavioral change (increased physical and social engagement in their communities) throughout the week.

SUMMARY:
This study will investigate the feasibility of a 6-month community walking program for people with Parkinson's disease (PD) and their care partners in greater Saint Louis, Missouri region. The walking program will consist of weekly, organized walking groups at the Missouri Botanical Gardens. Participants in the program will use Nordic walking poles during the walks. The walking group(s) will meet once per week and will be supervised by walking group leaders from Saint Louis University. Participants will be given a smart watch to wear that will help step counts will be tracked in real-time. The program is designed to get people with Parkinson's disease out of their homes, cultivate a culture of connection with others with Parkinson's disease, and to be collectively accountable for a common goal toward increasing their physical and social engagement in their communities.

ELIGIBILITY:
Inclusion Criteria:

* 30-85 years old
* Neurologist-diagnosed Parkinson's disease
* Able to walk independently with or without a walking aid (e.g., cane, walker)
* Willing to participate in study for at least 6 months

Exclusion Criteria:

* Health diagnosis that would limit exercise participation (e.g., heart problems, uncontrolled blood pressure, exercise-induced asthma).
* Additional neurologic disease or injury beyond Parkinson's disease.
* Evidence of significant cognitive impairment. This will be determined by completing the Montreal Cognitive Assessment
* Participants with poor walking ability (determined using the Timed Up and Go Test during initial testing).

Ages: 30 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2027-03-31 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Safety/Rate of Falls - Feasibility | From enrollment to both the 6 and 12 month endpoints
  The rate falls related to walking program participation.
Enrollment - Feasibility | Through enrollment of all the study participants
  The percentage of eligible participants that enroll in the study.
Attendance - Feasibility | Enrollment through the 6- and 12-month endpoints
  The percentage of attended walking program session across all enrolled participants.

SECONDARY OUTCOMES:
Steps per Day | From baseline assessment through the the end of the fall reporting period at 18 months
  This outcome will be captured via wearable sensors worn through the duration of study participation.
Balance Discordance | From baseline assessment through the 6- and 12-month endpoints
  This is the difference between actual balance confidence (captured via the activities specific balance confidence scale) and predicted balance confidence (modeled from time to complete the Timed Up and Go Test).
Loneliness | From baseline assessment through the 6- and 12-month endpoints
  Assessed with the 20 item UCLA loneliness scale in which subjects rate the degree of loneliness that they experience in daily life. The scale has a minimum score of 20 and maximum score of 80 with higher scores indicating that the individual is experience more loneliness.
Social Connection | From baseline assessment through the 6- and 12-month endpoints
  Assessed with the Berkman-Syme Social Network Index, an 11-item questionnaire in which participants rate their perceived social network and isolation. The index has a minimum score of zero and maximum score of 11 with higher score indicating a larger and stronger social network.

CONTACTS AND LOCATIONS:
Locations (1):
- Integrated Health and Movement Science Laboratory, Saint Louis University, St Louis, Missouri, United States